CLINICAL TRIAL: NCT02368548
Title: Randomized Clinical Trial of a Pharmaceutical Care Program in Chronic Patients Users of an Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Ana Juanes, Pharmacist, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IIBSP-PAF-2011-81; IIBSP-PAF-2011-81 (Other: Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau)
Record Dates: First submitted 2015-01-20; First posted 2015-02-23 (Estimated); Last update posted 2015-02-23 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure; Pulmonary Disease, Chronic Obstructive
Keywords: Pharmaceutical care; Emergency Service
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pharmaceutical care program (Experimental): 1. Initiated in the Emergency Department (ED):
     1. Review of home medication and medication reconciliation based on Primary Care data
     2. Patient interview. Assessment of the patient's knowledge on the pharmacological treatment
     3. Development of the pharmacological history and registration in the medical record
     4. Adequacy of drug therapy. Identification of Drug Related Problems including reconciliation errors (DRP) and communication to medical team
     5. Pharmacotherapy monitoring
     6. Treatment validation and medication reconciliation at discharge
  2. During the hospitalization (if admission from the ED):
     1. Treatment review and medication reconciliation
     2. Pharmacokinetics monitoring
     3. Retrospective validation of prescriptions and assessment of drugs appropriateness. DRP identification and communication to medical team
     4. Pharmacotherapy monitoring
     5. Validation and medication reconciliation at discharge
     6. Patient education at discharge
  Interventions: Other: Pharmaceutical Care Program
- Standard Care (Other): Stages:
  1. Pharmaceutical care program in the episode at the Emergency Department:
     a. There was no monitoring of the patient by the pharmacist. Retrospective validation of the prescriptions was not performed.
  2. During the hospitalization (if admission from the ED):
     1. Pharmacokinetics monitoring
     2. Retrospective validation of prescriptions and assessment of drugs appropriateness.
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Pharmaceutical Care Program — Intensive pharmaceutical care program, initiated in the emergency department, as described in its corresponding arm intervention description.
  Arms: Pharmaceutical care program
Other: Standard Care — Standard pharmaceutical care process, initiated at the hospital admission, as described in its corresponding arm intervention description.
  Arms: Standard Care

SUMMARY:
The study aims to assess the clinical and economic impact of a pharmaceutical care program initiated in the Emergency Department versus conventional follow-up of patients with decompensated heart failure/COPD.

DETAILED DESCRIPTION:
Clinical trial aimed to assess the impact of a pharmaceutical care program initiated in the Emergency Department vs standard care in patients with heart failure and/or COPD, conducted at the Hospital de la Santa Creu i Sant Pau (Barcelona, Spain) between Jan12-Feb13.

The researchers hypothesize that a systematic, standardized pharmaceutical care program may be related to a lower frequency of drug related problems (DRP). Moreover, the investigators also hypothesize that 6-month mortality, the average length of the hospital stay, and its related cost may also be decreased.

This study was approved by the Hospital de la Santa Creu i Sant Pau Ethics Committee. Written informed consent will be obtained from the participants .

The study will include 100 patients who fulfill all the inclusion criteria, described in the Eligibility Section.

ELIGIBILITY:
Inclusion Criteria:

* Age: 65 years and over
* Admission in the Emergency Department for a period equal to or higher than 12 hours;
* Number of home medication equal to or higher than four;
* Diagnose in the Emergency Department episode: decompensated heart failure and/or decompensated COPD.

Exclusion Criteria:

* Suffering from dementia, severe mental disorders and living in nursing homes.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Drug Related Problems (DRP) | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Patient health outcomes that are not consistent with the objectives of pharmacotherapy and are associated with the use or errors in the use of medicines
Mortality | 6-month after inclusion
  Patients who died during the following 6 months after inclusion
Average length of the hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Duration of the stay (in hours) from the emergency episode until discharge from the hospital
Readmissions | 6-month after inclusion
  Number of visits (emergency department/hospitalization) due to HF and/or COPD decompensation after the first episode (inclusion in the study), in the next 1180 days.
Average cost of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 10 days
  Average money spent per patient in Euros.

REFERENCES:
- [Background] Baena MI, Fajardo PC, Pintor-Marmol A, Faus MJ, Marin R, Zarzuelo A, Martinez-Olmos J, Martinez-Martinez F. Negative clinical outcomes of medication resulting in emergency department visits. Eur J Clin Pharmacol. 2014 Jan;70(1):79-87. doi: 10.1007/s00228-013-1562-0. Epub 2013 Oct 3. PMID 24091839
- [Background] Gorgas Torner MQ, Paez Vives F, Camos Ramio J, de Puig Cabrera E, Jolonch Santasusagna P, Homs Peipoch E, Schoenenberger Arnaiz JA, Codina Jane C, Gomez-Arbones J. [Integrated pharmaceutical care programme in patients with chronic diseases]. Farm Hosp. 2012 Jul-Aug;36(4):229-39. doi: 10.1016/j.farma.2011.06.015. Epub 2011 Dec 3. Spanish. PMID 22137609
- [Background] Gillespie U, Alassaad A, Henrohn D, Garmo H, Hammarlund-Udenaes M, Toss H, Kettis-Lindblad A, Melhus H, Morlin C. A comprehensive pharmacist intervention to reduce morbidity in patients 80 years or older: a randomized controlled trial. Arch Intern Med. 2009 May 11;169(9):894-900. doi: 10.1001/archinternmed.2009.71. PMID 19433702
- [Background] Koehler BE, Richter KM, Youngblood L, Cohen BA, Prengler ID, Cheng D, Masica AL. Reduction of 30-day postdischarge hospital readmission or emergency department (ED) visit rates in high-risk elderly medical patients through delivery of a targeted care bundle. J Hosp Med. 2009 Apr;4(4):211-8. doi: 10.1002/jhm.427. PMID 19388074
- [Background] Castro I, Guardiola JM, Tuneu L, Sala ML, Faus MJ, Mangues MA. Drug-related visits to the emergency department in a Spanish university hospital. Int J Clin Pharm. 2013 Oct;35(5):727-35. doi: 10.1007/s11096-013-9795-7. Epub 2013 May 22. PMID 23695594
- [Derived] Juanes A, Garin N, Mangues MA, Herrera S, Puig M, Faus MJ, Baena MI. Impact of a pharmaceutical care programme for patients with chronic disease initiated at the emergency department on drug-related negative outcomes: a randomised controlled trial. Eur J Hosp Pharm. 2018 Sep;25(5):274-280. doi: 10.1136/ejhpharm-2016-001055. Epub 2017 Feb 23. PMID 31157039
- See also: Third Consensus of Granada on Drug Related Problems (DRP) and Negative — http://farmacia.ugr.es/ars/pdf/374.pdf